CLINICAL TRIAL: NCT04347447
Title: Effect of Incorporating Lean Beef Into a Protein-rich Diet During Resistance Training Program on Skeletal Muscle and Connective Tissue Strength and Quality in Older Women
Brief Title: Effect of Incorporating Lean Beef Into a Protein-rich Diet During Resistance Training on Muscle and Tendon Strength in Older Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Purdue University (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Principal Investigator, Chad C. Carroll, Assistant Professor,Health and Kinesiology, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-2019-218
Record Dates: First submitted 2020-03-31; First posted 2020-04-15 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Sarcopenia; Aging
Keywords: women; beef; skeletal muscle; tendon; connective tissue; older adults
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: three intervention groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal protein diet (Experimental): The normal protein diet (Control) will contain the RDA for protein of (0.8 g/kg/d), with the protein provided from a variety of animal and plant-based sources, including lean beef (one 3-oz portion per week), chicken, eggs, dairy, beans, grains, nuts, seeds.
  Interventions: Other: Exercise training
- a beef protein-rich diet (Experimental): High protein diet predominantly provided from lean beef (one 3-oz portion per day; total beef intake 24 oz/week). The energy content of the additional protein foods will be isocalorically offset by substitution for low-protein foods.
  Interventions: Other: Exercise training
- a protein-rich diet non-red meat (Experimental): High-protein group from a variety of animal and plant-based sources (excluding additional red meats).
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — All groups will complete a supervised 12-week resistance training protocol, 3 days per week.

SUMMARY:
Loss of muscle mass and strength is a well-established outcome of normal aging. Muscle strength and mobility are also dependent on the quality and strength of connective tissue, which surrounds skeletal muscle. These layers, which are continuous with tendons, allow for the effective transfer of tension from skeletal muscle to bone to enable movement. Importantly, skeletal muscle strength is directly related to connective tissue strength. Greater tendon connective tissue cross-sectional area and stiffness optimize force transfer through tendon to maximize musculoskeletal function. As with skeletal muscle, tendon connective tissue quality declines with age. Previous research indicates that resistance training can improve muscle strength in older adults, but may not counter the effects of aging on tendon. The specific problem is that no approaches are available that benefit both skeletal muscle and tendon health to minimize loss of muscle mass and quality while also improving connective tissue quality and function in older adults. A critical need exists to assess approaches that improve both muscle and connective tissue strength and function. This need is highly relevant for older women, due to their higher risk of sarcopenia than men.

Resistance training, especially when combined with higher protein intake, has been consistently shown to improve muscle mass and strength in older adults. Further, emerging research indicates that diets rich in total and indispensable amino acids (as in beef) augment exercise-induced improvements in tendon cross-sectional area in rodents and young humans. However, limited research exists on the impact of beef consumption combined with resistance training on muscle and tendon tissue outcomes, especially in older women. This research study will assess the effects of consuming a healthy, protein-rich diet emphasizing lean beef, compared to a healthy, normal-protein, lower beef diet (control 1), and a healthy protein-rich, lower beef diet emphasizing non-beef/red meat protein (control 2) on resistance training-induced changes in muscle and tendon tissue size, strength, and quality in older women.

DETAILED DESCRIPTION:
Sarcopenia, i.e., loss of muscle mass and strength, is a well-established consequence of normal aging. Skeletal muscle strength and mobility is also dependent on the composition and mechanical properties of connective tissue, which encase skeletal muscle allowing for effective transfer of tension developed during cross-bridge cycling. Importantly, skeletal muscle strength and function is directly related to connective tissue strength. Specifically, greater tendon connective tissue cross-sectional area (CSA) and stiffness optimize force transfer through tendon to maximize musculoskeletal function, including muscle power output, locomotion economy, and control of balance. As with skeletal muscle, aging leads to the decline of tendon connective tissue quality, including reductions in tendon collagen (the primary structural component of tendon), and a decrease in tendon CSA. Previous research indicates that resistance training (RT) can improve muscle mass and strength in older adults but may not counter the effects of aging on tendon. Specifically, a 12-week RT protocol improved tendon properties in young but not older adults. The specific problem is that no approaches are available that target both skeletal muscle and tendon health to minimize loss of muscle mass and quality while simultaneously improving connective tissue quality and function in older adults. Therefore, a critical need exists to scientifically assess interventions that concomitantly improve muscle and connective tissue strength and function. This need is highly relevant for older women, due to their higher risk of sarcopenia than men.

Resistance training, especially when combined with higher protein intake, has been consistently shown to improve muscle mass and strength in older adults. However, limited research exists on the impact of beef consumption combined with RT on sarcopenia-related outcomes, especially in older women. Further, emerging research indicates that diets rich in leucine or glycine (as in beef) augment resistance or aerobic exercise-induced improvements in tendon CSA in rodents and young humans. However, the potential benefit of lean proteins, such as beef, on connective tissue adaptations in older adults requires investigation. This study will assess the effects of consuming a healthy, protein-rich diet emphasizing lean beef on RT-induced changes in skeletal muscle and tendon connective tissue size, strength, and quality in older women. It is hypothesized that consumption of a healthy diet high in protein from predominately lean beef will augment improvements in both skeletal muscle and tendon responses to RT, when compared to consuming a healthy diet with normal or high-protein and less total red meat. The overall healthy diet will be modeled from the U.S. Healthy Eating Pattern and consistent with the 2015-2020 Dietary Guidelines for Americans.

ELIGIBILITY:
Inclusion Criteria:

* Women 60-80 years old.
* BMI < 40
* Women with HbA1c less than 6.5% (non-diabetic)
* Must be able to complete upper and lower body resistance training exercise

Exclusion Criteria:

* Chronic users of analgesic medications such as acetaminophen, ibuprofen, or prescription cyclooxygenase inhibitors -Prisoners-
* Users of tobacco
* Individuals with claustrophobia or implanted objects who cannot complete on MRI scan
* Individuals with any orthopedic condition that would prevent them from properly performing exercise.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle Mass | within 1 week prior to beginning the intervention and then again within 1 week of completing the intervention
  MRI will be used to determine thigh muscle volume before and after the intervention
Tendon Connective Tissue Stiffness | within 1 week prior to beginning the intervention and then again within 1 week of completing the intervention
  Patellar tendon stiffness will be assessed using ultrasound methods
Skeletal Muscle Strength | within 1 week prior to beginning the intervention and then again within 1 week of completing the intervention
  Strength will be determined using the 1 repetition maximum method
Patellar Tendon Size | within 1 week prior to beginning the intervention and then again within 1 week of completing the intervention
  MRI will be used to determine tendon cross-sectional area and length

SECONDARY OUTCOMES:
Blood glucose | 6 and 12 weeks
  a blood sample will be taken for assessment of blood glucose
HbA1c | 6 and 12 weeks
  a blood sample will be taken for assessment of blood glucose
Cholesterol | 6 and 12 weeks
  a blood sample will be taken for assessment of cholesterol levels
Triglycerides | 6 and 12 weeks
  a blood sample will be taken for assessment of total triglyceride levels

CONTACTS AND LOCATIONS:
Overall Officials: Chad Carroll, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carroll CC, Campbell NW, Lewis RL, Preston SE, Garrett CM, Winstone HM, Barker AC, Vanos JM, Stouder LS, Reyes C, Fortino MA, Goergen CJ, Hass ZJ, Campbell WW. Greater Protein Intake Emphasizing Lean Beef Does Not Affect Resistance Training-Induced Adaptations in Skeletal Muscle and Tendon of Older Women: A Randomized Controlled Feeding Trial. J Nutr. 2024 Jun;154(6):1803-1814. doi: 10.1016/j.tjnut.2024.04.001. Epub 2024 Apr 9. PMID 38604504